CLINICAL TRIAL: NCT01791114
Title: The Effect of Brown Adipose Tissue Activation on Insulin Sensitivity in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Labros Sidossis, Ph.D., Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-193
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2019-01

CONDITIONS: Insulin Sensitivity; Obesity
Keywords: Insulin sensitivity; Diabetes Prevention; Obesity; Brown adipose tissue
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Propranolol; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cold water consumption (Experimental): Subjects will participate in two trials as part of this protocol: a) cold water (4 °C) consumption and b) tepid (36 °C) water consumption
  Interventions: Other: Cold water consumption; Other: Tepid water consumption
- Meal consumption (Experimental): Subjects will participate in two trials as part of this protocol: a) High calorie meal consumption and two weeks later b) no meal consumption.
  Interventions: Other: Thermoneutral Conditions; Other: Meal consumption
- Cold exposure (Experimental): Participants will complete three studies: a) cold exposure study (above their individually determined shivering threshold ~ 16°C); b) Cold exposure plus 0.5mg/kg up to 40mg propranolol at the beginning of the metabolic study and again after 4-6 hrs; c) thermoneutral conditions (26 - 28°C).
  Interventions: Other: Cold exposure; Other: Cold exposure plus propranolol; Other: Thermoneutral Conditions
- Exercise (Experimental): Subjects between 18 and 35 years old will be asked to participate in two trials: a) Exercise, i.e. four times for 10 min- at 85% VO2max (maximal oxygen consumption). with 15-min breaks between each bout b) and two weeks later rest.
  Interventions: Other: Thermoneutral Conditions; Other: Exercise

INTERVENTIONS:
Other: Cold exposure — For the cold exposure trial, the subjects will follow an individualized cold exposure protocol maximize the elicited non-shivering thermogenesis. Subjects will be wearing liquid conditioned garments (Polar Products Inc, Stow, OH). The temperature will initially be set at 18°C, then decreased at 1 degree celsius intervals thought the air- conditioned temperature control bath until subjects report shivering. Electromyography (EMG; Delsys, Bagnoli 8, Boston, MA) will be performed continuously to verify shivering muscle activity. Upon shivering, the temperature will be increased by 1degree Celsius intervals until shivering resides. Subjects' core temperature will be measured at 10-second intervals with the use of a telemetric pill (Core Temp Inc., Palmetto, FL).
  Arms: Cold exposure
Other: Cold exposure plus propranolol — For the cold exposure plus propanol trial, temperature will be titrated as previously described. The non-selective beta-adrenergic antagonist propranolol (0.5mg/kg and up to 40) will be given orally before the beginning of the study and again after 4-6 hours. In case participant's heart rate after propranolol administration decreases below 50 beats per min or systolic blood pressure below 90 mmHg second dose of propranolol will not be administered. Heart rate and blood pressure will be monitored continuously throughout the study. Propranolol doses up to 80 mg have been shown to significantly reduce fludeoxyglucose (FDG) uptake in brown fat in clinical patients.
  Arms: Cold exposure
Other: Thermoneutral Conditions — Subjects will be exposed to thermoneutral conditions (26 - 28°C)
  Arms: Cold exposure; Exercise; Meal consumption
Other: Cold water consumption — Subjects will be asked to consume cold water (4 °C,10 ml/ kg body weight within 10 minutes)
  Arms: Cold water consumption
Other: Tepid water consumption — Subjects will be asked to consume cold water (36 C,10 ml/ kg body weight within 10 minutes)
  Arms: Cold water consumption
Other: Exercise — Subject will be asked to complete four bouts of exercise for 10 min- at 85% of their maximal oxygen consumption (VO2max) with 15-min breaks between each bout
  Arms: Exercise
Other: Meal consumption — Subjects will be asked to consume a high calorie meal (12 kcal/kg, 50% carbohydrates, 30% fat, and 20% protein) within 15 minutes.
  Arms: Meal consumption

SUMMARY:
Recent findings document the presence of active brown adipose tissue (BAT) in humans. Cold exposure via adrenergic stimulation activates BAT, which combusts significant amounts of blood glucose and free fatty acid (FFA) to produce heat. Animal studies suggest that BAT activation improves insulin sensitivity. However, the effect of cold-induced BAT activation on insulin sensitivity and glucose kinetics in humans remains unknown. The investigators' central hypothesis is that cold-induced BAT activation increases whole body insulin sensitivity in humans via augmented plasma glucose and FFA clearance. The specific aims of this study are to define the effects of prolonged (8h) cold exposure BAT activation on: insulin sensitivity (Aim 1); lipolysis and plasma glucose and FFA kinetics (Aim 2); on thermoregulation (Aim 3). Moreover, the investigators plan to investigate for alternative ways, which can activate BAT including cold water ingestion, a single meal ingestion, and a single bout of moderate intensity exercise (Aim 4). For the cold exposure study, subjects will complete 3 trials: a) 8hrs of cold exposure at their individually determined shivering threshold; b) 8hrs of cold exposure at their individually determined shivering threshold plus propranolol; c) 8hrs in thermoneutral conditions (26 - 28°C). For the rest of the arms of subjects will complete two trials: cold or tepid water ingestion, a single meal ingestion or no food ingestion, and a single bout of moderate intensity exercise or no exercise.To study the above aims, the investigators will use positron emission tomography - computed tomography, hyperinsulinemic euglycemic clamp, infusion of stable isotopes, and tissue biopsies. The findings will illuminate the role of BAT on plasma substrate regulation and insulin sensitivity and may aid in the development of lifestyle recommendations and pharmacotherapy for the prevention and treatment of diabetes and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* men or women
* 18-75 years old
* BMI 20-40 kg/m2

Exclusion Criteria:

* taking diabetes medications
* liver/renal/endocrine/heart disease
* obstructive disease of the gastrointestinal tract
* impaired gag reflex or swallowing disorder
* history of GI surgery or fenilization of esophagus
* GI hypomotility disorder
* cancer
* thyroid or hormone replacement treatment
* beta-blockers
* anabolic or corticosteroids the last 6 mo
* pregnant/lactating women
* individuals that are likely to need PET/CT in the near future for medical reasons
* bleeding disorders/ anemia
* positive hepatitis or HIV screening
* weight less than 36 kg
* pacemaker or other implanted electromedical device
* alcohol and drug abuse
* tobacco use
* impaired cognition
* asthma
* chronic obstructive pulmonary disease (COPD) or other reactive airway diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | After 8hrs of cold exposure or thermoneutral conditions
  Insulin sensitivity will be measured using the euglycemic hyperinsulinemic insulin clamp method

SECONDARY OUTCOMES:
Metabolic profile | During the 8hr trial or on the following day
  Evaluation of metabolic profile will include measurement of various metabolites (glucose, triglycerides, very low-density (VLDL)-triglycerides, non-esterified fatty acids, lipoproteins, apo-B) and hormones (leptin, adiponectin, insulin, ghrelin).

OTHER OUTCOMES:
Substrate kinetics | During the 8hr study
  We will use a stable isotopes to assess substrate kinetics. Specifically, a primed, constant 4hr infusion of 6,6-D2-glucose to assess glucose kinetics; b) a constant 4hr infusion of potassium uniformly labelled with carbon 13 [U-13C16] palmitate to assess FFA kinetics (27, 28); and c) a primed, constant, 4hr infusion of [1,1,2,3,3-2H5]glycerol dissolved in 0.9% NaCl solution, to assess whole body lipolysis , and) a bolus of labeled with carbon13 sodium bicarbonate(NaHCO3) dissolved in 09% sodium chloride (NaCl) solution to assess substrate oxidation.
Thermoregulation | During the first 5-6 hrs of the cold exposure study
  We will use a telemetric pill and wireless thermistors to monitor the body core and skin temperatures of the participants. Moreover, thermal sensation will be assessed using a visual analog scale of the American Society of Heating, Refrigerating, and Air-Conditioning Engineers. Heart rate and blood pressure will be also measured to assess the cardiovascular response to cold exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Labros Sidossis, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch at Galveston, Galveston, Texas, United States

REFERENCES:
- [Derived] Chondronikola M, Volpi E, Borsheim E, Chao T, Porter C, Annamalai P, Yfanti C, Labbe SM, Hurren NM, Malagaris I, Cesani F, Sidossis LS. Brown Adipose Tissue Is Linked to a Distinct Thermoregulatory Response to Mild Cold in People. Front Physiol. 2016 Apr 19;7:129. doi: 10.3389/fphys.2016.00129. eCollection 2016. PMID 27148068
- [Derived] Chondronikola M, Volpi E, Borsheim E, Porter C, Annamalai P, Enerback S, Lidell ME, Saraf MK, Labbe SM, Hurren NM, Yfanti C, Chao T, Andersen CR, Cesani F, Hawkins H, Sidossis LS. Brown adipose tissue improves whole-body glucose homeostasis and insulin sensitivity in humans. Diabetes. 2014 Dec;63(12):4089-99. doi: 10.2337/db14-0746. Epub 2014 Jul 23. PMID 25056438